CLINICAL TRIAL: NCT05444881
Title: THE BYS COVID-19 COPING INTERVENTION STUDY- PHASE II: A RANDOMIZED CONTROLLED TRIAL OF AN mHEALTH MINDFULNESS PROGRAM
Brief Title: Boricua Youth Study COVID-19 Coping Intervention Study
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: U.S. Department of Health and Human Services OHRP issued an FWA restriction on NYSPI research that included a pause of human subjects research as of June 23, 2023. This study will resume recruitment after OHRP has approved the resumption of research.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Morgan Stanley Children's Hospital (Other)
Responsible Party: Principal Investigator, Cristiane Duarte, Ruane Professor for the Implementation of Science for Child and Adolescent mental Health (in Psychiatry) at CUMC, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB #8273
Record Dates: First submitted 2022-06-24; First posted 2022-07-06 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Psychological Stress; Depression; Anxiety
MeSH Terms: conditions — Stress, Psychological; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Parents will be randomly assigned to either receive treatment immediately after consent is obtained or wait for 6 weeks. Parents and children in the intervention group will be asked to complete a phone assessment at baseline and immediately after the intervention (posttreatment) to assess preliminary clinical outcomes. Hair and saliva samples will be collected from both parents and children at baseline and posttreatment. Parents will also complete a brief semi-structured interview on the feasibility and acceptability of the mHealth mindfulness program at posttreatment. There will be a brief follow-up phone assessment for clinical outcomes in parents at 4-8 weeks posttreatment. Parents and children in the waitlist group will complete the same measures as those in the intervention group at baseline and after their six weeks wait before they complete the mHealth intervention. There will be a brief phone assessment at posttreatment (parent and child) and 4-8 weeks follow-up (parent only).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 10-20 minutes a day of mindfulness meditation practice through the Headspace app.
  Participants will receive daily reminders to participate and receive weekly calls to assess adherence.
  Participants will be briefed on the telephone on how to use the app and receive recommendations of possible meditations they can engage with throughout the 6 weeks of participation.
  Interventions: Behavioral: Mindfulness-based Intervention (Headspace TM)
- Waitlist Control (No Intervention): Waitlist Control

INTERVENTIONS:
Behavioral: Mindfulness-based Intervention (Headspace TM) — A commercially available mindfulness mobile phone application (HeadspaceTM) will be used. The use of HeadspaceTM in the current protocol is approved by NYSPI Information Technology Services.
  An mHealth mindfulness program such as Headspace provides self-paced, guided mindfulness meditations through a website or mobile app (iOS and Android). The program consists of basic meditation courses as well as courses targeting stress management, anxiety, depression, and parenting. Based on the qualitative interviews with parents in Phase I, psychoeducation will be included on mindfulness practice and mental health, emphasizing basic meditation courses, and asking parents to complete daily assignments of 10 to 20 min a day during the 6-week period. As an engagement strategy, every week participants in the intervention group will receive a call or an email or text message (depends on preference; partisans may opt out to receive email/text messages).
  Arms: Intervention

SUMMARY:
The current study is the second phase of a two-part study to examine the feasibility and utility of using an mHealth mindfulness intervention to help parents mitigate the stress associated with the impact of sustained community crisis situations, such as COVID-19 and its consequences, on low-income families living in under-resourced settings.

DETAILED DESCRIPTION:
The current pilot study is a randomized controlled trial with an intervention (n=25 parent-child pairs) and a waitlist control (n=15 parent-child pairs) group that examines the feasibility, acceptability, and preliminary outcomes of the mHealth mindfulness program for parents. Parent participants will utilize a commercially available mobile phone application, Headspace TM, to complete 10-20 minutes of mindfulness exercises daily for six weeks. The investigators will measure the feasibility and acceptability of the mHealth mindfulness program for parents and clinical outcomes in both parents and children and also explore the effects of the intervention on stress markers including cortisol and inflammation (C-reactive protein (CRP) and Interleukin-6 (Il-6)).

Participants will recruit from an existing longitudinal cohort, the Boricua Youth Study (BYS; NYSPI IRB protocols #4187R and #6476) and BYS-ECHO (NYSPI IRB Protocols # 7377). The BYS is an epidemiological study on the development of psychiatric disorders in Puerto Rican children. Participants for the current study are a subsample G1 BYS participants who are parents of youth (G2) ages 3 to 12 years old.

Aim 1: To exam the feasibility and acceptability of an mHealth mindfulness program to reduce psychosocial distress among parents of children between 5 and 12 years old (N=40 parent-child pairs) Aim 2: To test preliminary clinical outcome for parents (psychosocial distress and functioning) and child (behavioral and emotional problems) Exploratory Aim: To explore the effects of an mHealth mindfulness-based intervention (MBI) on stress markers including cortisol and inflammation (CRP and IL-6)

Study procedure:

Intervention group:

* Screen
* Consent
* Randomization
* Baseline assessments for the parent (30 minutes including parent self-reports and parent reports of child) and child self-reports (15 minutes)
* 6-week Intervention with daily assignments (10-20 minutes per day)
* Posttreatment assessments for the parent (40 minutes including self-reports, parent report of child, and a brief exit interview) and child self-reports (15 minutes)
* 4-8 week posttreatment follow up assessments for the parent (5-10 minutes)

Waitlist group :

* Screen
* Consent
* Randomization
* Baseline assessments for the parent (30 minutes including parent self-reports and parent report of child) and child self-report (15 minutes)
* 6-week waitlist
* Post waitlist/Pretreatment for the parent (30 minutes including parent self-reports and parent report of child) and child self-report (15 minutes)
* 6-week Intervention with daily assignments (10-20 minutes per day)
* Posttreatment assessments for the parent (20-30 minutes including parent self-reports, parent report of child, and exit interview)
* 4-8 week posttreatment follow up assessments of parent self-reports (5-10 minutes)

ELIGIBILITY:
Inclusion Criteria:

1. BYS participants in the NY cohort
2. Have a child/children ages 3 to 12 years
3. access to a smartphone, tablet, or computer with at least periodic internet access

Exclusion Criteria:

1. Psychiatric risks (e.g., homicidally, suicidality including ideation and attempts, psychosis; answering "yes" to the PHQ-9 suicidal idea question, Q9)
2. Severe depressive symptoms (i.e., PHQ-9=20 or above)
3. Engagement of regular mindfulness, meditation, or yoga practice 3 or more times per week or enrollment in a mindfulness program

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale (PSS-10) | Baseline, Posttreatment (6 weeks), Follow up (10-14 weeks)
  Perceived Stress (10 items, rated 1-4, higher scores mean higher perceived stress)

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder-7 (GAD-7) | Baseline, Posttreatment (6 weeks), Follow up (10-14 weeks)
  Anxiety symptoms (7 items, rated 0-3, higher scores mean higher generalized anxiety symptoms)
Change in Patient Health Questionnaire-9 (PHQ-9) | Baseline, Posttreatment (6 weeks), Follow up (10-14 weeks)
  Depression Symptoms (9 items, rated 0-3, higher scores mean higher depressive symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane Duarte, PhD, Principal Investigator — New York State Psychiatric Institute; Tenneill Murray, MPH, Study Director — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No